CLINICAL TRIAL: NCT02800226
Title: Pilot Study Comparing 10Hz Repetitive Transcranial Magnetic Stimulation (rTMS) vs. Intermittent Theta Burst Stimulation (iTBS) for Treatment Resistant Depression
Brief Title: Pilot Study Comparing 10hz vs Theta Burst Stimulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-02340
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10Hz (Experimental): High Frequency Left repetitive transcranial magnetic stimulation five days per week for 4-6 weeks
  Interventions: Device: 10Hz
- iTBS (Active Comparator): intermittent Theta Burst Stimulation (iTBS) five days per week for 4-6 weeks
  Interventions: Device: iTBS

INTERVENTIONS:
Device: 10Hz — Magventure Cool B70 Coil with X100 Stimulator and ANT Neuronavigation System
  Arms: 10Hz
Device: iTBS — Magventure Cool B70 Coil with X100 Stimulator and ANT Neuronavigation System
  Arms: iTBS

SUMMARY:
This pilot study aims at exploring the efficacy of iTBS compared to 10Hz protocol and explore potential biomarkers of treatment response

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* voluntary and competent to consent
* Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of Major Depressive Disorder (MDD), single, recurrent between ages 18-65
* failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of ≥ 3 in the current episode or have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2)
* have a score of ≥ 18 on the Hamilton Depression Rating Score 17-item (HDRS-17)
* have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening able to adhere to the treatment schedule
* Pass the TMS adult safety screening (TASS) questionnaire
* have normal thyroid functioning based on pre-study blood work

Exclusion Criteria:

* have a history of substance dependence or abuse within the last 3 months
* have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* have active suicidal intent
* are pregnant
* have a lifetime MINI diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform, delusional disorder, or current psychotic symptoms
* have a MINI diagnosis of obsessive-compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia assessed by a study investigator to be primary and causing greater impairment than MDD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in the Hamilton Depression Rating scale 17-item (HDRS-17) score | baseline, 1, 4, and 12 weeks post-treatment
  A 50% improvement in the score is considered response to rTMS. A final score of <8 is categorized as remission.

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, Principal Investigator — University of British Columia
Locations (1):
- Non-Invasive Neurostimulation Therapies lab, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ge R, Downar J, Blumberger DM, Daskalakis ZJ, Vila-Rodriguez F. Functional connectivity of the anterior cingulate cortex predicts treatment outcome for rTMS in treatment-resistant depression at 3-month follow-up. Brain Stimul. 2020 Jan-Feb;13(1):206-214. doi: 10.1016/j.brs.2019.10.012. Epub 2019 Oct 18. PMID 31668646
- [Derived] Shalbaf R, Brenner C, Pang C, Blumberger DM, Downar J, Daskalakis ZJ, Tham J, Lam RW, Farzan F, Vila-Rodriguez F. Non-linear Entropy Analysis in EEG to Predict Treatment Response to Repetitive Transcranial Magnetic Stimulation in Depression. Front Pharmacol. 2018 Oct 30;9:1188. doi: 10.3389/fphar.2018.01188. eCollection 2018. PMID 30425640
- See also: Laboratory Website — http://NINET.CA